CLINICAL TRIAL: NCT04015505
Title: Does the Timeline Approach With Older Adults Experiencing Depression Reduce Negative Affect, and Result in Increased Self-compassion and Wisdom for Managing Current Difficulties? A Single Case Experimental Design
Brief Title: Can Life's Wisdom Help Counter Depression? Evaluating the CBT Timeline Approach for Older Adults With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 248358
Record Dates: First submitted 2019-06-17; First posted 2019-07-11 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Depression in Old Age
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Single case experimental design, with non-concurrent across-participants multiple baselines. All participants will receive the intervention, with a period of measured baseline stability acting as the control for each participant. Participants will not need to take part in the study simultaneously.
  Participants will be randomly allocated to one of three baseline conditions:
  Group A = 2 weeks baseline Group B = 3 weeks baseline Group C = 4 weeks baseline
  Following their baseline, each participant will complete a 5 week intervention period where they receive 5 sessions of the therapy. Throughout their baseline and intervention period, each participant will complete weekly measures of mood and a daily visual analogue scale. Each participant will also complete measures of self-compassion and wisdom at the start of baseline, end of baseline and end of intervention. Each participant will complete all measures again at one time point 1 month following the end of their intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will receive 5 sessions of a psychological (talking therapy) intervention based on the wisdom enhancement 'timeline technique' within cognitive behavioural therapy for older adults.
  Interventions: Behavioral: Cognitive Behavioural Therapy for older adults: wisdom enhancement 'timeline technique'

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for older adults: wisdom enhancement 'timeline technique' — The intervention is comprised of five one-hour sessions of structured talking therapy, where participants create a timeline of their life with significant events included. Through dialogue with the therapist and structured worksheets, participants are encouraged to reflect on events in their life to recognise and develop qualities of resilience and self-compassion. They are then asked to use 'the wisdom of their years' to develop strategies to manage difficulties they are currently facing. Participants will also be asked to complete worksheets and try out new strategies between sessions.

SUMMARY:
This study aims to evaluate a specific psychological technique to help older adults with depression improve their mood and develop or utilise their 'wisdom' for managing their current difficulties. The United Kingdom (UK) population is ageing and effective psychological therapies for older adults need to be well evaluated and developed. This study aims to develop evidence for this technique, and links between gerontological theories of wisdom and clinical psychology.

The 'timeline' technique (Laidlaw, 2010, 2015) is recommended within Cognitive Behavioural Therapy (CBT) for older adults. CBT is the most evidenced based psychological treatment for a range of psychiatric disorders including depression. Outcome studies have found that older people are just as likely to respond to CBT as younger people.

This technique draws on theories of 'wisdom', where one's wisdom can develop from how they reflect on their life experiences. Depressed individuals may view their lives in overgeneralised negative ways, making this process harder. The timeline technique asks people to create a timeline of their lives. Through reflection and discussion of past events, they are helped to recognise personal resilience, develop self-compassion, and utilise their wisdom for managing current difficulties. This technique requires specific evaluation to determine its validity and effectiveness.

This study uses a single-case experimental research design to allow conclusions to be drawn from a small number of participants. Six individuals from primary and secondary care mental health waiting lists, as well as third sector providers, aged over 60 and experiencing depression or low mood, will be invited to take part in a short testing of this technique. Individuals will be asked to measure their mood and complete relevant questionnaires throughout their involvement in the study and will do this for up to 4 weeks on their own. They will then meet with a trainee clinical psychologist for five weekly sessions of a structured therapy using the timeline technique.

DETAILED DESCRIPTION:
BACKGROUND

The United Kingdom (UK) population is getting older, with those over 65 predicted to reach 24% by 2037 (Office for National Statistics, 2017). With improved quality of life and advances in healthcare, there is increased pressure on services to cater for the wellbeing of older adults. UK government states that depression affects one in five older people living in the community (UK Government, 2017). Depression is therefore a significant mental health condition for older adults and for which effective treatments and approaches are required. As such, there is a growing need to tailor psychological therapies to the older adult population and for new techniques to be well evaluated.

'Cognitive behavioural therapy (CBT) for older adults' augments traditional evidence-based CBT for the older adult population with 'age-appropriate' techniques, developed from lifespan developmental models and gerontological theory to help enhance treatment outcomes for older adults (Knight & Laidlaw, 2009; Laidlaw, 2010). One technique is the 'wisdom enhancement' timeline technique (Laidlaw, 2010, 2015; Laidlaw & Kishita, 2015), which builds on a psychological model of wisdom applied to clinical psychology. The technique has roots in classical cognitive behavioural techniques but is distinctive in how it uses one's life narrative as a resource. The timeline technique can be regarded as an innovative and structured way of using peoples' life narratives and experiences in a cognitive-behavioural framework to evolve the psychological resource of wisdom and increase mood and coping in the present. It is time-limited and present problem focused. The timeline technique is recommended in Increased Access to Psychological Therapies Services (IAPT) guidelines for CBT for older adults, meaning that it will be routinely used in National Health Service (NHS) settings in England. The timeline technique is theorised to improve mood by increasing self-acceptance and wisdom. However, the technique has not been specifically tested in detail.

PURPOSE OF THE STUDY

This study will investigate in detail the 'wisdom enhancement' timeline technique for helping older adults with depression develop 'wisdom', self-compassion and improve mood. The study will use a single-case experimental design to evaluate the technique's effectiveness and mechanisms of change. It will provide a valuable examination of a specific recommended CBT technique, where there is a general need for more testing of individual components of therapy. The results from this investigation will help inform further developments of wisdom enhancement models in clinical psychology and efficacy of CBT for older adults.

RESEARCH AIM

The primary aim of this study is to evaluate the 'timeline technique' (Laidlaw, 2015) with older adults experiencing mild-moderate depression. This will be achieved by delivering a short psychological intervention to older adults using the timeline technique, based on appropriate guidelines. Principle research questions:

1. Does the timeline intervention reduce negative affect?
2. Does the timeline intervention increase self-compassion?
3. Does the timeline intervention increase wisdom for managing current difficulties?

STUDY DESIGN

This study uses a single case experimental design (SCED) to measure the effects that the 'timeline' intervention has on mood, self-compassion and wisdom, as measured by structured self-report questionnaires and idiographic measures. Older adults experiencing depression/low mood will be recruited from NHS primary and secondary care or third sector psychological treatment waiting lists.

SCEDs have long been used in psychology intervention research and are a useful method for examining the effectiveness of an intervention on individuals with only a few participants (Morgan & Morgan, 2001; Kazdin, 2011). Unlike randomised controlled trials, each participant acts as their own control by measuring their baseline state for a period of time before the intervention is introduced. Each participant will take part in three phases:

1. Baseline phase: participants will complete weekly standardised measures of mood and daily idiographic measures of mood, self-compassion and wisdom.
2. Intervention phase: participants will receive a 5 week psychological intervention, whilst continuing to complete the baseline measures. This will allow for any observable change in mood during the onset of the intervention to be determined.
3. Participants will complete a single set of follow up measures 1 month after the intervention phase ends.

Participants will also complete standardised measures of mood, self-compassion and wisdom at pre-baseline, pre-intervention and post-intervention time points, to allow for further between phase testing. Measurement during the intervention phase and at follow up will account for effects of the intervention that accrue slowly over time and test if any effects are sustained.

The study adopts an across-participant multiple baseline component which means that each participant will be randomly assigned to one of three pre-determined baseline phases of differing lengths:

Group A: 2 weeks Group B: 3 weeks Group C: 4 weeks The multiple baseline design is the most frequent design used in psychology single case studies (Smith, 2012) and allows for greater control for determining when changes in the target variable are attributed to a specific study phase.

Participants will take part once they are recruited and it is convenient for them to take part, rather than needing to all start simultaneously. This is therefore considered a non-concurrent multiple baseline design and allows greater flexibility for both researchers and participants.

ADDITIONAL INFO

This study is taking place as part of the chief investigator's research training and qualification for a UK Doctorate in Clinical Psychology.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 60.
* Primary problem depression, as measured by the screening tool PHQ-9 cut off point of 5.
* Currently on a waiting list for psychological treatment or considered treatment resistant.
* Low risk for suicide or self-harm, as screened through recruiting clinicians, health records and clinical judgement of the researcher
* Absence of cognitive impairment or substance misuse
* Participants should be on a stable dose, at least 3 months without change, of antidepressant medication
* Able to speak and understand English

Exclusion Criteria:

* Must not already be receiving any active psychological treatment for depression, or changes to any antidepressant medication in the past three months. If participants are on antidepressant medication which has not been changed in the last three months they will be still be eligible - this will be considered a stable dose.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
9-item Patient Health Questionnaire - assessing levels of change over time for each participant | Group A: Weekly throughout study completion, up to 7 weeks and once at 1 month follow-up: at week 11
  9 item self-report measure for depression. (PHQ-9; Kroenke, Spitzer, & Williams, 2001).
  The PHQ-9 is a brief and widely used nine-item self-report tool for measuring depression. Total scores range from 0 to 27 with higher scores suggesting higher severity of depression. This measure will be used as a primary outcome measure to monitor changes in mood across the duration of the study and will be assessed each week. The PHQ-9 will also be used as a study screening tool with a score above 5 (indicating mild depression; Kroenke et al., 2001) set as the cut-off point.
9-item Patient Health Questionnaire - assessing levels of change over time for each participant | Group B: Weekly throughout study completion, up to 8 weeks and once at 1 month follow-up: at week 12
  9 item self-report measure for depression. (PHQ-9; Kroenke, Spitzer, & Williams, 2001).
  The PHQ-9 is a brief and widely used nine-item self-report tool for measuring depression. Total scores range from 0 to 27 with higher scores suggesting higher severity of depression. This measure will be used as a primary outcome measure to monitor changes in mood across the duration of the study and will be assessed each week. The PHQ-9 will also be used as a study screening tool with a score above 5 (indicating mild depression; Kroenke et al., 2001) set as the cut-off point.
9-item Patient Health Questionnaire - assessing levels of change over time for each participant | Group C: Weekly throughout study completion, up to 9 weeks and once at 1 month follow-up: at week 13
  9 item self-report measure for depression. (PHQ-9; Kroenke, Spitzer, & Williams, 2001).
  The PHQ-9 is a brief and widely used nine-item self-report tool for measuring depression. Total scores range from 0 to 27 with higher scores suggesting higher severity of depression. This measure will be used as a primary outcome measure to monitor changes in mood across the duration of the study and will be assessed each week. The PHQ-9 will also be used as a study screening tool with a score above 5 (indicating mild depression; Kroenke et al., 2001) set as the cut-off point.
10-item Geriatric Anxiety Scale - assessing levels of change over time for each participant | Group A: Weekly throughout study completion, up to 7 weeks and once at 1 month follow-up: at week 11
  10 item self-report measure for anxiety in later life. (GAS-10; Mueller et al, 2015).
  The GAS-10 is a brief 10 item scale is a shorty form scale adapted from the 30-item Geriatric Anxiety Scale (Segal, June, Payne, Coolidge, & Yochim, 2010). It is a self-report questionnaire designed to measure severity of anxiety for older adults. Total scores range from 0 to 30, with higher total scores meaning higher levels of anxiety.
10-item Geriatric Anxiety Scale - assessing levels of change over time for each participant | Group B: Weekly throughout study completion, up to 8 weeks and once at 1 month follow-up: at week 12
  10 item self-report measure for anxiety in later life. (GAS-10; Mueller et al, 2015).
  The GAS-10 is a brief 10 item scale is a shorty form scale adapted from the 30-item Geriatric Anxiety Scale (Segal, June, Payne, Coolidge, & Yochim, 2010). It is a self-report questionnaire designed to measure severity of anxiety for older adults. Total scores range from 0 to 30, with higher total scores meaning higher levels of anxiety.
10-item Geriatric Anxiety Scale - assessing levels of change over time for each participant | Group C: Weekly throughout study completion, up to 9 weeks and once at 1 month follow-up: at week 13
  10 item self-report measure for anxiety in later life. (GAS-10; Mueller et al, 2015).
  The GAS-10 is a brief 10 item scale is a shorty form scale adapted from the 30-item Geriatric Anxiety Scale (Segal, June, Payne, Coolidge, & Yochim, 2010). It is a self-report questionnaire designed to measure severity of anxiety for older adults. Total scores range from 0 to 30, with higher total scores meaning higher levels of anxiety.
Idiographic visual analogue scale - assessing daily change over time for each participant | Group A: Daily through study completion, for total of 43 days and once at 1 month following end of intervention period: at week 11
  Self-reported idiographic visual analogue scale with specific questions developed in accordance with the study hypotheses:
  1. Today, I feel that my mood is good
  2. Today, I feel accepting of myself
  3. Today, I feel that I can use the wisdom of my life to help deal with current difficulties
  Idiographic measures are often used as well as standardized measures in single case design. They allow for specific target constructs to be measured in a way that is repeatable and efficient. The visual analogue scale consists of a ten-centimeter line anchored at either end with maximal and minimal extremes of the dimension being measured. Participants put a mark on the line, with the mark closer to the right side indicating stronger agreement of that statement. A numerical measurement of the line gives a score for each statement based on length (between 0 and 10.)
Idiographic visual analogue scale - assessing daily change over time for each participant | Group B: Daily through study completion, for total of 50 days and once at 1 month following end of intervention period: at week 12
  Self-reported idiographic visual analogue scale with specific questions developed in accordance with the study hypotheses:
  1. Today, I feel that my mood is good
  2. Today, I feel accepting of myself
  3. Today, I feel that I can use the wisdom of my life to help deal with current difficulties
  Idiographic measures are often used as well as standardized measures in single case design. They allow for specific target constructs to be measured in a way that is repeatable and efficient. The visual analogue scale consists of a ten-centimeter line anchored at either end with maximal and minimal extremes of the dimension being measured. Participants put a mark on the line, with the mark closer to the right side indicating stronger agreement of that statement. A numerical measurement of the line gives a score for each statement based on length (between 0 and 10.)
Idiographic visual analogue scale - assessing daily change over time for each participant | Group C: Daily through study completion, for total of 57 days and once at 1 month following end of intervention period: at week 13
  Self-reported idiographic visual analogue scale with specific questions developed in accordance with the study hypotheses:
  1. Today, I feel that my mood is good
  2. Today, I feel accepting of myself
  3. Today, I feel that I can use the wisdom of my life to help deal with current difficulties
  Idiographic measures are often used as well as standardized measures in single case design. They allow for specific target constructs to be measured in a way that is repeatable and efficient. The visual analogue scale consists of a ten-centimeter line anchored at either end with maximal and minimal extremes of the dimension being measured. Participants put a mark on the line, with the mark closer to the right side indicating stronger agreement of that statement. A numerical measurement of the line gives a score for each statement based on length (between 0 and 10.)
Self-compassion scale - assessing levels of change over time for each participant | Group A: At week 1, week 3, week 7, week 11.
  26-item self-report measure of self-compassion (SCS; Neff, 2003)
  26-item self-report measure of self-compassion measures overall self-compassion as well as six subscales, representing components of self-compassion: self-kindness versus self-judgment, sense of common humanity versus isolation, and mindfulness versus over-identification. Responses to each question are given on a 5-point Likert scale, from 'almost never' to 'almost always'. Subscale scores are computed by calculating the mean of subscale item responses, and therefore range from 0-5 with higher scores indicating higher levels of that construct. Total self-compassion score is calculated by reverse scoring the negative subscale items before calculating subscale means - self-judgment, isolation, and over-identification, then calculating a grand mean of all six subscale means. The total score ranges from 0-5 with higher scores indicating higher levels overall self-compassion.
Self-compassion scale - assessing levels of change over time for each participant | Group B: At week 1, week 4, week 8, week 12.
  26-item self-report measure of self-compassion (SCS; Neff, 2003)
  26-item self-report measure of self-compassion measures overall self-compassion as well as six subscales, representing components of self-compassion: self-kindness versus self-judgment, sense of common humanity versus isolation, and mindfulness versus over-identification. Responses to each question are given on a 5-point Likert scale, from 'almost never' to 'almost always'. Subscale scores are computed by calculating the mean of subscale item responses, and therefore range from 0-5 with higher scores indicating higher levels of that construct. Total self-compassion score is calculated by reverse scoring the negative subscale items before calculating subscale means - self-judgment, isolation, and over-identification, then calculating a grand mean of all six subscale means. The total score ranges from 0-5 with higher scores indicating higher levels overall self-compassion.
Self-compassion scale - assessing levels of change over time for each participant | Group C: At week 1, week 5, week, 9, week 13
  26-item self-report measure of self-compassion (SCS; Neff, 2003)
  26-item self-report measure of self-compassion measures overall self-compassion as well as six subscales, representing components of self-compassion: self-kindness versus self-judgment, sense of common humanity versus isolation, and mindfulness versus over-identification. Responses to each question are given on a 5-point Likert scale, from 'almost never' to 'almost always'. Subscale scores are computed by calculating the mean of subscale item responses, and therefore range from 0-5 with higher scores indicating higher levels of that construct. Total self-compassion score is calculated by reverse scoring the negative subscale items before calculating subscale means - self-judgment, isolation, and over-identification, then calculating a grand mean of all six subscale means. The total score ranges from 0-5 with higher scores indicating higher levels overall self-compassion.
Self-Assessed Wisdom Scale (SAWS) - assessing levels of change over time for each participant | Group A: At week 1, week 3, week 7, week 11.
  40-item self-report measure of wisdom (SAWS; Webster, 2007)
  This 40-item self-report measure of wisdom uses a 6-point Likert scale to measure five subscales of wisdom: critical life experience, reminiscence and reflectiveness, openness, emotional regulation, and humor.
  Each subsale total ranges from 0 to 40, with higher numbers indicating higher levels of that construct.
  Adding total subscale scores together will generate a total SAWS wisdom score, with values ranging from 40 to 200, with a higher score indicating an overall higher level of wisdom.
Self-Assessed Wisdom Scale (SAWS) - assessing levels of change over time for each participant | Group B: At week 1, week 4, week 8, week 12.
  40-item self-report measure of wisdom (SAWS; Webster, 2007)
  This 40-item self-report measure of wisdom uses a 6-point Likert scale to measure five subscales of wisdom: critical life experience, reminiscence and reflectiveness, openness, emotional regulation, and humor.
  Each subsale total ranges from 0 to 40, with higher numbers indicating higher levels of that construct.
  Adding total subscale scores together will generate a total SAWS wisdom score, with values ranging from 40 to 200, with a higher score indicating an overall higher level of wisdom.
Self-Assessed Wisdom Scale (SAWS) - assessing levels of change over time for each participant | Group C: At week 1, week 5, week, 9, week 13
  40-item self-report measure of wisdom (SAWS; Webster, 2007)
  This 40-item self-report measure of wisdom uses a 6-point Likert scale to measure five subscales of wisdom: critical life experience, reminiscence and reflectiveness, openness, emotional regulation, and humor.
  Each subsale total ranges from 0 to 40, with higher numbers indicating higher levels of that construct.
  Adding total subscale scores together will generate a total SAWS wisdom score, with values ranging from 40 to 200, with a higher score indicating an overall higher level of wisdom.

OTHER OUTCOMES:
Change interview questionnaire (non standardised brief qualitative questionnaire) | Group A: At week 7 / End of intervention period
  The 'Change interview questionnaire' is a three question qualitative questionnaire that has been created by the research team to be used specifically for this study. It is therefore not a standardised measure or scale.
  The questionnaire comprises of three qualitative questions based on the key information elicited in the semi-structured 'Change Interview' (Elliot, 2002), adapted to the format of a written questionnaire.
  This questionnaire asks the following three questions:
  1. What has changed for you over the course of the study?
  2. Why do you think these changes occurred?
  3. What has been helpful?
  Participants are asked to write qualitative answers to each question using the free space provided after each question.
  The answers to these questions will not be included in any formal analysis but will provide additional information in helping to evaluate the validity of any intervention effects for each case.
Change interview questionnaire (non standardised brief qualitative questionnaire) | Group B: At week 8 / End of intervention period
  The 'Change interview questionnaire' is a three question qualitative questionnaire that has been created by the research team to be used specifically for this study. It is therefore not a standardised measure or scale.
  The questionnaire comprises of three qualitative questions based on the key information elicited in the semi-structured 'Change Interview' (Elliot, 2002), adapted to the format of a written questionnaire.
  This questionnaire asks the following three questions:
  1. What has changed for you over the course of the study?
  2. Why do you think these changes occurred?
  3. What has been helpful?
  Participants are asked to write qualitative answers to each question using the free space provided after each question.
  The answers to these questions will not be included in any formal analysis but will provide additional information in helping to evaluate the validity of any intervention effects for each case.
Change interview questionnaire (non standardised brief qualitative questionnaire) | Group C: At week 9 / End of intervention period
  The 'Change interview questionnaire' is a three question qualitative questionnaire that has been created by the research team to be used specifically for this study. It is therefore not a standardised measure or scale.
  The questionnaire comprises of three qualitative questions based on the key information elicited in the semi-structured 'Change Interview' (Elliot, 2002), adapted to the format of a written questionnaire.
  This questionnaire asks the following three questions:
  1. What has changed for you over the course of the study?
  2. Why do you think these changes occurred?
  3. What has been helpful?
  Participants are asked to write qualitative answers to each question using the free space provided after each question.
  The answers to these questions will not be included in any formal analysis but will provide additional information in helping to evaluate the validity of any intervention effects for each case.

CONTACTS AND LOCATIONS:
Overall Officials: Adam JZ Kadri, Principal Investigator — University of East Anglia
Locations (2):
- United Kingdom (2):
  - Cambridge and Peterborough NHS Foundation Trust, Cambridge
  - Norfolk and Suffolk NHS Foundation Trust, Norwich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kazdin, AE. Single-case research designs: Methods for clinical and applied settings. Oxford University Press, 2011.
- [Background] Knight BG, Laidlaw, K. Translational theory: A wisdom-based model for psychological interventions to enhance well-being in later life. In V. L. Bengston, D. Gans, N. M. Pulney, & M. Silverstein (Eds.), Handbook of theories of aging (pp. 693-705). New York, NY, US: Springer Publishing Co. 2009.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Laidlaw K. Are attitudes to ageing and wisdom enhancement legitimate targets for CBT for late life depression and anxiety?. Nordic Psychology 62: 27-42, 2010.
- [Background] Laidlaw K. Enhancing cognitive behavior therapy with older people using gerontological theories as vehicles for change. Casebook of Clinical Geropsychology: International Perspectives on Practice, 17, 2010.
- [Background] Laidlaw K, Kishita, N. Age-appropriate augmented cognitive behavior therapy to enhance treatment outcome for late-life depression and anxiety disorders. Geropsych 28: 57-66, 2015.
- [Background] Laidlaw K. CBT for older people: An introduction. Sage, London, 2015.
- [Background] Morgan DL, Morgan RK. Single-participant research design. Bringing science to managed care. Am Psychol. 2001 Feb;56(2):119-27. PMID 11279805
- [Background] Mueller AE, Segal DL, Gavett B, Marty MA, Yochim B, June A, Coolidge FL. Geriatric Anxiety Scale: item response theory analysis, differential item functioning, and creation of a ten-item short form (GAS-10). Int Psychogeriatr. 2015 Jul;27(7):1099-111. doi: 10.1017/S1041610214000210. Epub 2014 Feb 27. PMID 24576589
- [Background] Neff KD. The development and validation of a scale to measure self-compassion. Self and identity 2(3): 223-250, 2003.
- [Background] Office for National Statistics (2017). Overview of the UK population: July 2017. Retrieved from https://www.ons.gov.uk/peoplepopulationandcommunity/populationandmigration/populationestimates/articles/overviewoftheukpopulation/july2017
- [Background] Smith JD. Single-case experimental designs: a systematic review of published research and current standards. Psychol Methods. 2012 Dec;17(4):510-50. doi: 10.1037/a0029312. Epub 2012 Jul 30. PMID 22845874
- [Background] Webster JD. Measuring the character strength of wisdom. Int J Aging Hum Dev. 2007;65(2):163-83. doi: 10.2190/AG.65.2.d. PMID 17957986
- [Background] UK Government (2017) Living Well in Older Years. Retrieved from: https://www.gov.uk/government/publications/better-mental-health-jsna-toolkit/7-living-well-in-older-years#fn:4
- [Background] Elliott R. Hermeneutic single-case efficacy design. Psychother Res. 2002 Mar 1;12(1):1-21. doi: 10.1080/713869614. PMID 22471329